CLINICAL TRIAL: NCT04658563
Title: The Effect of High Density Hatha Yoga Training on Physical Fitness, Respiratory Functions and Quality of Life in Healthy Adolescents
Brief Title: Yoga for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Neslihan Duruturk, Associated Proffesor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA18 / 345
Record Dates: First submitted 2020-10-22; First posted 2020-12-08 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Yoga
Keywords: Yoga; physical fitness; adolescent; quality of life; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Yoga (Experimental): High-density HY training; average 90-110 minutes, 2 sessions per week under the supervision of the physiotherapist, once a week as a home program, will be applied for a total of 8 weeks to the first group.
  Interventions: Other: High Density Exercise Training Program - Yoga
- Group 2: Control (No Intervention): Individuals in the second group will not included in any exercise training program

INTERVENTIONS:
Other: High Density Exercise Training Program - Yoga — A total of 8 weeks will be applied in our study, each session of the high-density yoga program will be started with 10 minute pranayama (breath) exercises as it is in classical yoga as a preliminary preparation for the participation of individuals; the program will be completed by applying 10-20 minutes warming-stretching movements, 40 minutes surya namaskar (SN) sets, 20-30 minutes dynamic yoga asanas and 10 minutes savasana. Participants will be encouraged to study the perceived difficulty levels between 14 and 17 using the Borg scale during the sessions
  Other Names: Yoga
  Arms: Group 1: Yoga

SUMMARY:
Purpose: Specific effects of high-density Hatha Yoga(HY) training in adolescents have not yet been clarified. Aim of our study is to investigate the effects of high-density HY education on physical fitness, pulmonary function and quality of life in healthy adolescents. Methods: 28 female adolescents will be randomly divided into two groups as yoga training and control groups. Training group will receive high-density HY training for 8 weeks, two days a week under the supervision of a physiotherapist and one day a week home program. Control group will not receive any exercise. Flexibility of individuals will be determined by sit-reach, back scratching, lateral flexion tests; muscular endurance by sit-ups, sit down-stand up on chair tests, balance by time up-go test; cardiorespiratory capacity by incremental shuttle walking test(ISWT) and respiratory functions by spirometry, quality of life will be determined by with the Quality of Life Scale for Children.

ELIGIBILITY:
Inclusion Criteria:

- Female adolescents between the ages of 14 and 18

Exclusion Criteria:

- Individuals with recent muscular skeletal, neuromuscular and chronic systemic diseases that could prevent exercise

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Health-Related Physical Fitness - Upper extremity flexibility | 8 weeks
  Lateral Flexion and Back Scratch Tests will be performed to evaluate upper extremity flexibility.
Assessment of Health-Related Physical Fitness - Lower extremity flexibility | 8 weeks
  Sit and Reach Test will be performed to assess lower extremity flexibility.
Assessment of Health-Related Physical Fitness - Balance | 8 weeks
  Time up-go test will be performed to evaluate the balance levels of the patients.
Assessment of Health-Related Physical Fitness - Endurance | 8 weeks
  Upper extremity muscular endurance will be evaluated by Sit-up Test and lower extremity muscular endurance by Sit up-down on Chair Test
Cardiorespiratory endurance | 8 weeks
  Incremental Shuttle Walking Test: The test is controlled by audible warnings between two marked points, 9 meters apart; individuals will be asked to walk at increasing speed with stimulus, and each meter they walk will be recorded as a shuttle.
Assessment of Respiratory Functions | 8 weeks
  The pulmonary functions of the individuals will be evaluated in the sitting position using the portable spirometer device (COSMED, Micro Quark Spirometer, Rome, Italy) according to the ATS/ERS criteria. The individuals who participated in the study will be informed about the test before the test. The test will be repeated twice and the best results will be recorded. The individual is seated on a chair without a cuff, a latch is attached to his nose, his mouth is asked to be closed tightly so that the edges of the mouths could fully grasp the device. In respiratory function test, forced vital capacity (FVC) (Liter-L and %), first-second forced expiratory volume (FEV1)(L and %), FEV1/FVC, peak flow rate (PEF)(L/second), 25-75% of forced expiratory flow rate (FEF (25-75%)(L)), inspiratory capacity (IC) (L) and vital capasity (VC) (L) values will be recorded along with expected values and percentages by age, height, body weight and gender.
Forced vital capacity (FVC) | 8 weeks
  Forced vital capacity (FVC) will be measured in Liter and %.
First-second forced expiratory volume (FEV1) | 8 weeks
  First-second forced expiratory volume (FEV1) will be measured in Liter and %.
Peak flow rate (PEF) | 8 weeks
  Peak flow rate (PEF) will be measured in Liter/second.
25-75% of forced expiratory flow rate (FEF (25-75%) | 8 weeks
  25-75% of forced expiratory flow rate will be measured in Liter.
Inspiratory capacity (IC) | 8 weeks
  Inspiratory capacity (IC) will be measured in Liter.
Vital capacity (VC) | 8 weeks
  Vital capacity (VC) will be measured in Liter.
Assessment of quality of life | 8 weeks
  The form which is prepared for adolescents aged 13-18 and validated and reliable in our country of The Pediatric Quality of Life Inventory. The 23 items of the scale developed for children aged 2-18 are scored between 0-100; the answers will be 100 if 'never' are preferred, 75 if 'rarely, 50 if 'sometimes, 25 if 'often, and 0 if 'always,. The higher the total score, the better the quality of life is.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No